CLINICAL TRIAL: NCT06718348
Title: Assessing the Japet.W+ Lumbar Traction Device in Rehabilitation for Patients With Non-specific Mechanical Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grand Hôpital de Charleroi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EXO-Exoskeleton Japet.W
Record Dates: First submitted 2024-11-17; First posted 2024-12-05 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group CTRL (No Intervention): Participants will undergo 30 sessions of conventional physiotherapy
- Group EXP (Experimental): Participants will undergo 30 sessions of physiotherapy with the use of the Japet.W+ Exoskeleton
  Interventions: Other: Use of the Exoskeleton JAPET.W

INTERVENTIONS:
Other: Use of the Exoskeleton JAPET.W — Phsysiotherapy sessions with the support of the Exoskeleton JAPET.W
  Arms: Group EXP

SUMMARY:
The study will include patients suffering from nonspecific mechanical low back pain for more than 6 weeks. Two groups will be compared. A Control group and an Experimental group with the exoskeleton JAPET.W

DETAILED DESCRIPTION:
The study will include patients suffering from nonspecific mechanical low back pain for more than 6 weeks. The study will consist of two groups: a control group (Group CTRL) and an experimental group (Group EXP). Participants will be categorized into two categories: "workers," patients on temporary work leave due to low back pain, and "non-workers," patients unable to work due to this condition after exhausting all available therapeutic solutions.

Monitoring period (30 physiotherapy sessions): evaluations will be conducted at sessions 1, 15 and 30, on the two groups. Evaluation session 3 months after the end of the physiotherapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific mechanical low back pain for more than 6 weeks,
* 18 years ≤ Age < 80 years,
* Patient affiliated to the health social security system,
* Patient able to understand the information relating to the study and to sign the informed consent form

Exclusion Criteria:

* Specific low back pain (infectious, inflammatory, tumorous, or traumatic origin),
* Motor neurological deficits (peripheral or central),
* Extrapyramidal syndrome,
* Treatment with implanted neurostimulation,
* Cardiac or circulatory diseases or serious respiratory problems,
* Previous recent arthrodesis or recent lumbar prosthesis surgery,
* Surgery for herniated disc (<3 months),
* Fracture of the dorsolumbar spine or rib (<3 months),
* Skin lesions, contusions and stretching injuries of the trunk,
* Pregnancy,
* Individuals not tolerating the JAPET.W+ device during an initial trial,
* Under guardianship, curatorship or legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the efficacy of the JAPET.W - measurement of pain | Up to six months
  VAS scale for pain (o -no pain to 10 - pain as bad as it could possibly be) : rate of the patients who had at least -20 points/100 on the VAS for pain
Assessment of the efficacy of the JAPET.W - consumption of analgesic | Up to six months
  Assessment of analgesic use in the two groups at the first and last session
Assessment of the efficacy of the JAPET.W - functional assessment | Up to six months
  Mobility assessment with the french version of Oswestry Disablility Index. The scale goes from 0 - no pain to 5 - worse.
Assessment of the efficacy of the JAPET.W - Assessment of the kinesiophobia | Up to six months
  Comparison of the difference in TAMPA scale. This scale goes to 1-strongly disagree to 4-strongly agree with the proposal
Assessment of the efficacy of the JAPET.W - Assessment in quality of life | Up to six months
  Assessment in quality of life with EQ-5D-5L. The scale goes to 1-totally able to carry out the activity up to 5-totally unable to do so.
Assessment of the efficacy of the JAPET.W - Assessment of the Anxiety level | Up to six months
  Assessment of the Anxiety level with Hospital Anxiety Depression Scale. This scale ranges from 0-no anxiety to 3-totally anxious.

SECONDARY OUTCOMES:
Assessment of the safety of the JAPET.W | Up to six months
  Rate of patients who had at least one device related adverse event during the clinical investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Serge TROUSSEL, MD, Principal Investigator — Grand Hôpital de Charleroi
Locations (1):
- Grand Hôpital de Charleroi, Charleroi, Hainaut, Belgium

IPD SHARING:
Plan to Share IPD: No